CLINICAL TRIAL: NCT05617521
Title: Use of Abdominal Binder in Colonoscopies Performed by Trainees in Gastrointestinal Endoscopy: A Randomized, Double-blind, Sham-controlled Trial
Brief Title: Abdominal Binder in Colonoscopies Performed by Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Central Norte PEMEX (Other)
Responsible Party: Principal Investigator, Antonio Marmolejo, Principal investigator, Hospital Central Norte PEMEX
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DCAS-SSS GSM-HCN-INV-0043-2022
Record Dates: First submitted 2022-09-15; First posted 2022-11-15 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Performance of Colonoscopy; Tolerance of Colonoscopy
Keywords: abdominal binder; colonoscopy; looping

STUDY DESIGN:
Intervention Model Description: Once enrolled, patients will be randomized to either the abdominal binder (AB) group or the sham binder (SB) group in a 1:1 ratio.
Who Masked: Participant, Investigator
Masking Description: Randomization will be performed using a web-based computer system (Research Randomizer, Geoffrey C. Urbaniak and Scott Plous) by an independent statistician who had no other intervention in the study. An independent operator will print the randomization number and group for each participant (either the AB or SB group) in individual cards, which will be hidden in a locked black box by the same independent operator. Only the nurse, who will fit the abdominal binder to all the patients in a private space, will have access to the cards. Randomized data and cards will be concealed to study coordinators, endoscopists, clinical staff, and participants.
  For the participants in the SB group the same binder will be fitted, but once the patient is sedated, it will be loosened by the same nurse. The participants will wear a non-transparent gown over the binder so that it will not be visible to the endoscopists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Binder Intervention Group (Experimental): Patients randomized to the Abdominal Binder Intervention Group will have the abdominal binder (Revive 3-in-1 Postpartum Recovery Support Belt) secured firmly between the subcostal border and the anterior superior iliac spine area to the abdomen just prior the colonoscopy.
  Interventions: Device: Abdominal binder (Revive 3-in-1 Postpartum Recovery Support Belt)
- Sham Group (Sham Comparator): Sham Group will have the abdominal binder (Revive 3-in-1 Postpartum Recovery Support Belt) secured firmly between the subcostal border and the anterior superior iliac spine area to the abdomen just prior the colonoscopy but it will be loosened just prior the procedure.
  Interventions: Device: Loose abdominal binder (Revive 3-in-1 Postpartum Recovery Support Belt)

INTERVENTIONS:
Device: Abdominal binder (Revive 3-in-1 Postpartum Recovery Support Belt) — Revive 3-in-1 Postpartum Recovery Support Belt (KeaBabies® Co., CA, USA). An abdominal binder is a kind of elastic abdominal compression device
  Other Names: Revive 3-in-1 Postpartum Recovery Support Belt (KeaBabies® Co., CA, USA); Revive 3-in-1 abdominal binder
  Arms: Abdominal Binder Intervention Group
Device: Loose abdominal binder (Revive 3-in-1 Postpartum Recovery Support Belt) — Revive 3-in-1 Postpartum Recovery Support Belt (KeaBabies® Co., CA, USA). An abdominal binder is a kind of elastic abdominal compression device. It will be loosened just prior the procedure.
  Other Names: Revive 3-in-1 Postpartum Recovery Support Belt (KeaBabies® Co., CA, USA); Revive 3-in-1 abdominal binder
  Arms: Sham Group

SUMMARY:
This randomized trial will be conducted to evaluate the effectiveness and safety of an abdominal binder use during colonoscopy performed by gastrointestinal endoscopy fellow trainees. The investigators hypothesized that the abdominal binder use would facilitate and increase the effectiveness of the colonoscopy for inexperienced operators.

DETAILED DESCRIPTION:
It will be a randomized, double-blind, sham-controlled study. The trial will be performed at a single-center, Hospital Central Norte PEMEX, a tertiary center with a gastrointestinal endoscopy fellow trainee program with more than 10 years of experience. This trial will be conducted in accordance with the most recent version of the Declaration of Helsinki. The trial has been approved by the local ethical committee and research committee with the number DCAS-SSS GSM-HCN-INV-0043-2022. Written informed consent will be obtained from all the patients before participation. This manuscript will be reported in accordance with CONSORT guidelines.

Prior to the procedure, age, sex, height, weight, waist circumference (WC), body mass index (BMI), and colonoscopy indication of all participants will be recorded. Once enrolled, patients will be randomized to either the abdominal binder (AB) group or the sham binder (SB) group in a 1:1 ratio. Randomization will be performed using a web-based computer system (Research Randomizer, Geoffrey C. Urbaniak and Scott Plous) by an independent statistician who had no other intervention in the study. An independent operator will print the randomization number and group for each participant (either the AB or SB group) in individual cards, which will be hidden in a locked black box by the same independent operator. Only the nurse, who will fit the abdominal binder to all the patients in a private space, will have access to the cards. Randomized data and cards will be concealed to study coordinators, endoscopists, clinical staff, and participants.

The abdominal binder to be used for the patients allocated in the AB group was the Revive 3-in-1 Postpartum Recovery Support Belt (KeaBabies® Co., CA, USA). Its price is $29.96. The device is manufactured in two sizes, One Size and X-Large. For the patients with a waist circumference >110 cm it will be used the X-Large model. The three belts that make up the binder will be fitted to all the participants. Once placed, the binder will be adjusted to be located between the subcostal border and the anterior superior iliac spine. The participants will be asked to confirm that the binder is fastened tightly but not uncomfortably. For the participants in the SB group the same binder will be fitted, but once the patient is sedated, it will be loosened by the same nurse. The participants will wear a non-transparent gown over the binder so that it will not be visible to the endoscopists.

Bowel preparation with 4 L of polyethylene glycol solution in split-dose (2 L in the afternoon of the day before and 5 h before the colonoscopy) will be used in all the participants. In this trial, all colonoscopy procedures will be performed by two second-year fellow trainees in gastrointestinal endoscopy.

A standard video-colonoscope (EC-3890Li, PENTAX Co., Tokyo, Japan) will be used. All the patients will be placed in the left lateral decubitus position. Manual abdominal compression and postural change will be conducted by a technician when required by the endoscopy trainee or the attending endoscopist. Endoscopist or anesthesiology will be allowed to remove the binder at any time during the procedure if they resolve it was necessary for safety. Air insufflation will be used during colonoscopy.

Sample size was estimated over the primary outcome of the study based on pre-experimental data estimation and previously reported CIT and SD of similar studies with fellows' participation. It was calculated that 142 participants were needed to detect a 60-second difference in CIT (SD 110 sec), with 90% power and two-side alpha 0.05. Moreover, it was also calculated based on the frequency of ancillary maneuvers, using pre-experimental data estimation and literature data. It was found that 186 participants (93 per group) were needed to detect a 20% reduction in the use of ancillary maneuvers, with 90% power and two-side alpha 0.05. As a preventive measure in case of withdrawal or exclusion, the sample was expanded by 10%, a total of 206 patients, 103 in each group were included in the study.

Descriptive statistical analysis, including mean, mode, and frequencies will be performed for the description of the study data. The comparative analysis of the quantitative data will be previously subjected to normality evaluation by the Shapiro-Wilk test and graphical analyses. According to the normality, data comparative analysis will be performed either with a two-way Student's test or U Mann-Whitney test. For the comparative analyses of the categorical data (e.g., manual abdominal compression, postural change, need for intervention by the attending endoscopist) will be used chi-square or Fisher' exact test. A p value of <0.05 will be accepted as statistical significance. Statistical inferential analysis will be performed using RStudio® (R Core Team v.1.2.5033; R Foundation for Statistical Computing, Vienna, Austria) and SPSS® Statistics for Windows Version 23.0 (IBM Corp., Armonk, NY, USA). RStudio® (R Core Team v.1.2.5033) will be also used for drawing graphics. The study biostatistician (SA) will be blinded to the randomization phase and recollection data process.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults between the ages of 20-80
* Participants with ASA I-III (American Society of Anesthesiologists Class)
* Undergoing a colonoscopy at any of the study locations for:

I. CRC screening (first colonoscopy or 10 years follow up of negative exam). II. Surveillance (prior colonoscopy with polyps). III. Diagnostic colonoscopy performed to evaluate symptoms such as abdominal pain or rectal bleeding.

- Participants must have completed the full prescribed colonoscopy purgative preparation prior to their procedure and describe adequate cleansing.

Exclusion Criteria:

* Inability to provide informed consent.
* Patients with known or suspected pregnancy.
* Patients undergoing multiple procedures (e.g., upper and lower endoscopy).
* Previous colon resection surgery.
* History of problems with sedation or anesthesia.
* Patients with known or suspected diagnosis of inflammatory bowel disease (ulcerative colitis or Crohn's disease).
* Patients with a history of colorectal cancer or other intra-abdominal malignancy.
* Patients with open or recent wounds or skin rash on the anterior abdominal wall.
* History of cirrhosis or ascites.
* Patients who are medically unstable (American Society of Anesthesiology Class IV or above).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Arellano, M.D, Study Chair — Ethical committee president of the Hospital Central Norte PEMEX
Locations (1):
- Antonio Marmolejo, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: Formal requests for IPD information should be made by email (dr.marmolejo.ch@gmail.com) to the principal investigator Antonio Marmolejo

REFERENCES:
- [Background] Rex DK, Schoenfeld PS, Cohen J, Pike IM, Adler DG, Fennerty MB, Lieb JG 2nd, Park WG, Rizk MK, Sawhney MS, Shaheen NJ, Wani S, Weinberg DS. Quality indicators for colonoscopy. Gastrointest Endosc. 2015 Jan;81(1):31-53. doi: 10.1016/j.gie.2014.07.058. Epub 2014 Dec 2. No abstract available. PMID 25480100
- [Background] Toyoshima O, Nishizawa T, Sakitani K, Yamakawa T, Yoshida S, Fukagawa K, Hata K, Ishihara S, Suzuki H. Colonoscopy using back brace support belt: A randomized, prospective trial. JGH Open. 2019 Nov 7;4(3):441-445. doi: 10.1002/jgh3.12276. eCollection 2020 Jun. PMID 32514451
- [Background] Crockett SD, Cirri HO, Kelapure R, Galanko JA, Martin CF, Dellon ES. Use of an Abdominal Compression Device in Colonoscopy: A Randomized, Sham-Controlled Trial. Clin Gastroenterol Hepatol. 2016 Jun;14(6):850-857.e3. doi: 10.1016/j.cgh.2015.12.039. Epub 2016 Jan 6. PMID 26767313

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Started | 105 | 106
Completed | 105 | 106
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abdominal Binder Intervention Group | Sham Group | Total
Number analyzed (Participants) | 105 | 106 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.36 (11.98) | 65.33 (12.34) | 64.35 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 67 | 129
  Male | 43 | 39 | 82
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 105 | 106 | 211
Body Mass Index (IBM) [Median (Inter-Quartile Range); unit: kg/m^2] | 29 [25.7 to 32.2] | 27.4 [24 to 30.3] | 28.4 [24.7 to 31.6]
Height [Mean (Standard Deviation); unit: meter] | 1.64 (0.09) | 1.64 (0.07) | 1.64 (0.08)
Weight [Mean (Standard Deviation); unit: kilogram] | 78.44 (15.93) | 74.42 (13.92) | 76.42 (15.05)

OUTCOME MEASURES:

1. Primary Outcome: Mean Cecal Intubation Time
Description: Cecal intubation time will be defined as the time from insertion of the colonoscope into the rectum to identification of the base of the cecum
Time Frame: During colonoscopy, from insertion of scope into rectum to point in time when base of the cecum is identified, an average of 30 minutes.
Population: 8 participants with incomplete colonoscopy were excluded from the primary outcome analysis (intervention group n 4, sham group n 4).
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 101 | 102
second | 728 [544 to 902] | 774 [662 to 961]
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Superiority — Sample size was assessed over the primary outcome of the study based on pre-experimental data estimation. It was calculated that 142 participants were needed to detect a 60-second difference in CIT, with 90% power and two-side alpha 0.05. It was found that 186 participants were needed to detect a 20% reduction in the use of ancillary maneuvers. As a preventive measure in case of withdrawal or exclusion, the sample was expanded by 10%, a total of 206 patients; p = 0.008, Wilcoxon (Mann-Whitney) — The comparative analysis of the CIT was previously subjected to normality evaluation by the Shapiro-Wilk test. According to the rejection of normal distribution, comparative data analysis has been performed with a two-way Mann-Whitney U test

2. Secondary Outcome: Frequency of Use of Abdominal Pressure
Description: Binary data indicating individually when the abdominal pressure was used during the insertion phase of the procedure will be recorded.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 105 | 106
Participants | 15 | 58
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Chi-squared — For the comparison of abdominal pressure, Pearson chi-square test was used. The statistical significance level was accepted as p <0.05

3. Secondary Outcome: Length of Cecal Intubation
Description: The length of the colonoscope required to reach de cecum from the anus will be measured.
Time Frame: as for outcome 1
Population: Participants with incomplete colonoscopy were excluded from two of the main secondary outcomes (CIL and IVIT).
Measure: Median (Inter-Quartile Range); unit: centimeter
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 101 | 102
centimeter | 95 [90 to 100] | 100 [95 to 115]
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The comparative analysis of the CIL was previously subjected to normality evaluation by the Shapiro-Wilk test. According to the rejection of normal distribution, comparative data analysis has been performed with a two-way Mann-Whitney U test

4. Secondary Outcome: Frequency of Intervention by the Attending Endoscopist
Description: Binary data indicating individually if intervention by the attending endoscopist was required during the insertion phase of the procedure will be recorded.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 105 | 106
Participants | 6 | 11
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Superiority; p = 0.321, Chi-squared

5. Secondary Outcome: Colonoscopy Completion Rate
Description: Dichotomous outcome indicating if the procedure was complete.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 105 | 106
Participants | 100 | 102
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Superiority; p = 0.75, Fisher Exact

6. Secondary Outcome: Number of Participants With Mild, Moderate, and Severe Procedural Difficulty as Assessed by Trainees
Description: Immediately following completion of procedure, the study assistant will obtain the trainee's assessment of procedural difficulty according to three grades of severity: mild, moderate, and severe.
  *We found the 5-point scale more difficult to use in the dynamic of the endoscopy room. The Operator's Assessment of Procedural Difficulty scale was not used. The difficulty was rated as mild when the colonoscope was smoothly inserted, moderate when there were some difficulties quickly solved (less than 60 seconds), and severe when the difficulties were more difficult requiring a longer time (more than 60 seconds).
Time Frame: Immediately following completion of procedure when scope is removed from rectum, an average of 10 minutes after completion of the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 105 | 106
Participants
  Mild | 61 | 64
  Moderate | 38 | 23
  Severe | 6 | 19
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Superiority; p = 0.005, Chi-squared

7. Secondary Outcome: Number of Participants According to Colonoscopy Findings
Description: Findings such as polyps, cancer, diverticulum, and IBD (inflammatory bowel disease) detected during colonoscopy will be recorded.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 105 | 106
Participants
  Polyps | 36 | 30
  Diverticulosis | 42 | 44
  Colon Cancer | 0 | 1
  IBD | 1 | 0
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Other; p = 0.8, Fisher Exact

8. Secondary Outcome: Operator Perception of Patient Discomfort
Description: Immediately following completion of procedure, the study assistant will obtain operator's perception of patient discomfort during procedure according to the Gloucester score. The Gloucester score will be used. It is a comfort grading scale ranging from 1 to 5 points, with 1 point if no discomfort is present during the colonoscopy and 5 if there is extreme discomfort during the colonoscopy.
Time Frame: as for outcome 6
Population: We found the use of the Gloucester score difficult and subjective to use in the clinical scenario. The operators rated the episodes of discomfort in different ways, showing since the beginning a lack of consistency. The operator perception of patient discomfort was not evaluated. The data of this outcome were not collected for any patient.
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Additional Analgesic Drug Required to Complete Procedure
Description: Whether the patient needs an additional dose of analgesic drug to complete the colonoscopy.
Time Frame: During colonoscopy, from time point of insertion of scope into de rectum to point in time when scope is removed from rectum, an average of 30 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 105 | 106
Participants | 0 | 4
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Superiority; p = 0.12, Fisher Exact

10. Secondary Outcome: Patient Pain at Discharge
Description: The study assistant will interview patient just prior to discharge and obtain responses for pain according to a 10-point visual analog scale. The Visual analogue scale (VAS) will be used. It is a pain grading scale ranging from 0 to 10 points, with 0 if no pain and 10 if worst pain possible.
Time Frame: At single time point occurring after the colonoscopy, just prior to the patient being discharged from facility, an average of 90 minutes after completion of the procedure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 105 | 106
score on a scale | 2.22 (0.89) | 3.58 (0.88)
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Patient Satisfaction at Discharge
Description: The study assistant will interview patient just prior to discharge and obtain responses for satisfaction according to a 5-point Likert scale. The Satisfaction Likert scale will be used. It is a satisfaction grading scale ranging from 1 to 5 points, with 1 if very poor satisfaction and 5 if excellent satisfaction.
Time Frame: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 105 | 106
score on a scale | 3.65 (0.78) | 3.05 (0.88)
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Frequency of Use of Position Change
Description: Binary data indicating when the patient position change was used during the insertion phase of the procedure will be recorded.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 105 | 106
Participants | 2 | 12
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.01, Chi-squared — For the comparison of position change, Pearson chi-square test was used. The statistical significance level was accepted as p <0.05

13. Secondary Outcome: Additional Anesthetic Drug Required to Complete Procedure
Description: Whether the patient needs an additional dose of anesthetic drug to complete the colonoscopy.
Time Frame: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 105 | 106
Participants | 0 | 0
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Superiority; p = 1, Fisher Exact

ADVERSE EVENTS:
Time Frame: Time from the start of the sedation until the patient's discharge, approximately 2 hours
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Abdominal Binder Intervention Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/106
Other Adverse Events (participants affected / at risk) | 0/105 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT05617521/Prot_001.pdf
  • Statistical Analysis Plan (2023-09-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT05617521/SAP_002.pdf